CLINICAL TRIAL: NCT04631679
Title: Investigation of the Wash-out Effect of Intravenous Iron by Cell Savers
Brief Title: Investigation of the Wash-out Effect of Intravenous Iron by Cell Savers (WASH-OUT)
Acronym: WASH-OUT
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Collaborators: University of Muenster, Institute of Inorganic and Analytical Chemistry (Unknown)
Responsible Party: Sponsor
Other Study IDs: 09-Antl-19
Record Dates: First submitted 2020-11-10; First posted 2020-11-17 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Anemia; Anemia, Iron Deficiency; Iron Deficiency Anemia Treatment
Keywords: Anemia; Cell Saver; Iron Deficiency Anemia; Intravenous Iron; Ferric Carboxymaltose; Wash Out
MeSH Terms: conditions — Anemia; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Seven probes of patient's blood/serum, Cell Saver compounds or heart-lung machine are collected for each participant in Li-Heparin tubes (S-Monovette® 7,5ml Li-Heparin, Sarstedt AG & Co. KG, Nümbrecht, Germany) to examine ferric carboxymaltose levels in samples from different locations and time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: anemic patients with iron treatment: For Group A anemic patients (hemoglobin levels below 13g/dL in men and 12g/dL in women) with iron deficiency (transferrin saturation below 20% or ferritin serum level below 300μg/L) are screened in the Anesthesia pre-assessment clinic 1-4 days prior to cardiosurgical procedure (valve repair/implementation, aortocoronary bypass or a combination of both) and are treated with a single intravenous dose of 500 milligrams of ferric carboxymaltose in 100ml 0,9% sodium chloride solution as iron supplementation directly (FerInject® 50 mg/ml, 10 ml, Vifor Pharma Group, Switzerland).
- Group B: non-anemic patients without iron treatment: For Group B, non-anemic patients (hemoglobin levels above 13g/dL in men and 12g/dL in women) without iron deficiency (transferrin saturation above 20%, ferritin serum levels above 300μg/L) are screened in the Anesthesia pre-assessment clinic 1-4 days prior to cardiosurgical procedure (valve repair/implementation, aortocoronary bypass or both combined) and are not treated with iron supplementation.

SUMMARY:
The study is a pilot study, which involves cardiothoracic patients. Patients, who are scheduled for elective cardiosurgical procedure, will be seen in multidisciplinary anesthesia/Patient Blood Management (PBM) clinic and screened for anemia prior to surgery. Anemic patients will eventually be treated with 500mg of ferric carboxymaltose 1 to 4 days prior to surgery. A high blood loss is expected in these procedures (>500ml). Blood is collected and re-transfused to the patient via use of cell savers/ autologous blood restoration. The investigators will examine how fast intravenous ferric carboxymaltose is stored within the iron storage cells of the body, and how much remains within the patients blood at the time point of surgery. Next, the investigators will assess the wash out effect of iron via cell salvage. The hypothesis of this trial is that ferric carboxymaltose is washed out of the collected patient's blood by cell caver usage (Wash-Out Effect).

DETAILED DESCRIPTION:
Because of the short time frame between iron therapy to procedure in cardiac surgery due to the need to perform cardiac revascularization, the investigators aim to investigate how much of the iron compound ferric carboxymaltose is being stored within the iron storage cells of the human body, and how much remains in the patient's own blood at the time point of surgery. The terminal elimination half-life time of ferric carboxymaltose is known to be approximately 7.1 to 12.1 hours, with peak serum ferritin levels at 48h to 120h after administration. When high blood loss in a surgical procedure is expected, such as in cardiosurgical procedures, the usage of autologous cell salvage, so called "Cell Saver", is considered standard, good practice. The blood that is lost during surgery is collected and after a specified blood separation wash, being retransfused in form of concentrated red blood cells.

This trial aims to examine whether Cell Saver usage might recover high molecular iron complexes such as ferric carboxymaltose lost by bleeding intraoperatively or wash out these molecules.

If amount of lost blood during surgery is too low, that Cell Saver usage would not be possible otherwise, averagely 300ml of blood from the heart-lung machine are added to the cell saver to enable the process of cell saver use.

For each participant, 7 samples will be taken. The samples include patient's blood samples and samples from cell saver compartments (Washing solution, concentrates) as well as from the heart-lung-machine, in detail:

1. arterial patient's blood, preoperative, day of procedure, prior to surgery
2. blood from the heart-lung machine, intraoperative 30 minutes prior to end of use of the heart-lung machine, day of procedure
3. Cell Saver: washed-out compounds, intraoperative, after end of use of heart-lung machine, day of procedure
4. Cell Saver: produced red blood cell concentrate, intra- or postoperative, after end of use of heart-lung machine, day of procedure
5. arterial patient's blood, postoperative, day of procedure
6. venous patient's blood, 3. day postoperative
7. venous patient's blood, 7. day postoperative

By liquid chromatography inductively coupled plasma mass spectrometry (LC-ICP-MS) levels of ferric carboxymaltose are examined

1. in the patient's blood prior to surgery to determine the amount of ferric carboxymaltose within the patients blood prior to surgery, and after a certain time after the intravenous Infusion of ferric carboxymaltose (12-96 hours).
2. pre- and postoperatively and in cell saver compartments. If ferric carboxymaltose is detected in the washing solution of the Cell Saver System and not within the stored red blood cell concentrate, ferric carboxymaltose is washed out by the cell saver.

ELIGIBILITY:
Inclusion Criteria:

* scheduled cardiosurgical procedure such as valve surgery, aortocoronary bypass or both combined within 1-4 days after anesthesiological/PBM clinic
* for Group A: diagnosed anemia (hemoglobin levels below 13g/dL in men and 12g/dL in women) and iron-deficiency (transferrin saturation below 20% or ferritin serum level below 300μg/L), treatment with 500mg of ferric carboxymaltose (FerInject® 50 mg/ml, 10 ml, Vifor Pharma Group, Switzerland).

Exclusion Criteria:

* contraindication for intravenous iron therapy: severe infections, hepatocellular carcinoma, liver metastases, acute severe asthma, a simultaneous oral iron medication, another intravenous iron preparation, iron overload, chronic renal failure with regular intravenous iron substitution during dialysis treatment, age ≤18 years, pregnancy, lactation and being allergic to iron
* elevated C-reactive protein (CRP) and leukocyte levels (cut-off level for leucocytes for men was <10.9x10^3/μl and for women <12.68x10^3/μl, respectively)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of twenty-three patients undergoing elective cardiosurgical procedures (valve surgery, aortocoronary bypass or both combined) at University Hospital of Münster, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2019-11-08 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Ferric Carboxymaltose levels (µg/mL) | day of surgery to seven days after surgery
  Ferric Carboxymaltose levels in samples withdrawn from patient's blood, red blood cell concentrate of Cell Saver, heart-lung machine and washing solution prior to and after surgical procedure (µg/mL-Ferric carboxymaltose/plasma volume)

SECONDARY OUTCOMES:
Donor red blood cell concentrates | Beginning till end of surgery
  Additional substitution of donor red blood cell concentrates
Ferritin (ng/ml) | prior to intravenous iron supplementation
  Ferritin levels before intravenous iron supplementation
Ferritin (ng/ml) | point of intravenous iron supplementation until surgery
  Ferritin levels after intravenous iron supplementation
Ferritin (ng/ml) | 3 days after surgery
  Ferritin levels after intravenous iron supplementation
Ferritin (ng/ml) | 7 days after surgery
  Ferritin levels after intravenous iron supplementation
Hemoglobin levels (mg/dl) | prior to intravenous iron supplementation, 1 to 4 days prior to surgery
  Delta Hemoglobin levels between prior to IV iron substitution until surgery
Hemoglobin levels (mg/dl) | 3 days after surgery
  Hemoglobin levels after surgery
Hemoglobin levels (mg/dl) | 7 days after surgery
  Hemoglobin levels after surgery
Intraoperative blood loss (ml) | Beginning till end of surgery
  Blood volume lost while surgical procedure
Blood volume balance (ml) | Beginning till end of surgery
  Delta of intraoperatively given (infusions, transfusions) and lost (bleeding, withdrawn from heart-lung machine) volumes

CONTACTS AND LOCATIONS:
Overall Officials: Andrea U Steinbicker, MD, MPH, Study Chair — Dept. of Anesthesiology, Intensive Care and Pain Medicine, University Hospital of Münster
Locations (1):
- Dept. of Anesthesiology, Intensive Care and Pain Medicine, UKM, Münster, Germany

REFERENCES:
- [Derived] Olivier RMR, Macke M, Muller JC, Schrader L, Eveslage M, Rauer M, Wempe C, Martens S, Zarbock A, Wagner NM, Karst U, Dogan DY, Steinbicker AU. Perioperative Tracking of Intravenous Iron in Patients Undergoing On-Pump Cardiac Surgery: A Prospective, Single-Center Pilot Trial. Anesth Analg. 2023 Mar 1;136(3):578-587. doi: 10.1213/ANE.0000000000006372. Epub 2023 Feb 17. PMID 36811991